CLINICAL TRIAL: NCT01774838
Title: Vasoactive and Anti-inflammatory Effects of Prasugrel in Acute Coronary Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Tanja Rudolph, Consultant, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-1649
Record Dates: First submitted 2013-01-16; First posted 2013-01-24 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental): 3 months treatment with 10 mg prasugrel
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): 3 months treatment with clopidogrel 75 mg
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — 3 months treatment
  Other Names: Efient
  Arms: Prasugrel
Drug: Clopidogrel — 3 months treatment
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
To test the vasoactive and anti-inflammatory effects of prasugrel in patients with acute coronary syndrome endothelial function -as a surrogate parameter of NO bioavailability- and different markers of inflammation, oxidative stress and platelet activation will be assessed in patients with unstable angina.

DETAILED DESCRIPTION:
Trial Objectives To test the vasoactive and anti-inflammatory effects of prasugrel in patients with acute coronary syndrome, endothelial function -as a surrogate parameter of NO bioavailability- and different markers of inflammation, oxidative stress and platelet activation will be assessed in patients with unstable angina.

Trial Design Single center, double blind, double-dummy, randomized, parallel trial.

Endpoints

Primary Endpoint Assessment of endothelial function (FMD) via high-resolution ultrasound (Sonoline G50, 12 MHz linear array transducer, Siemens, Germany) by experienced sonographer.

Secondary Endpoints

* Non-invasive assessment of microvascular perfusion and oxygen saturation by laser Doppler perfusion imaging and tissue spectrometry (O2C, Lea Medizintechnik, Giessen, Germany)
* Determination of leukocyte activity: plasma MPO levels (ELISA), plasma elastase levels (ELISA)
* Assessment of platelet activity: plasma levels of sCD40 ligand (ELISA), RANTES (ELISA)
* Measurement of different oxidative stress markers: hsCRP (ELISA), CD40 ligand (ELISA), carbonylated proteins (ELISA), urinary 8-iso-PGF2α (gas chromatography mass spectrometry)
* Determination of platelet-leukocyte aggregates by fluorescent activated cell sorter (FACS)
* Assessment of platelet function (PADA-test)

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome, unstable angina
* planned percutaneous coronary intervention
* Written informed consent

Exclusion Criteria:

* - Age < 18 years or ≥75 years
* Body weight < 60 kg
* STEMI, NSTEMI
* Cardiogenic shock at the time of randomization
* Refractory ventricular arrhythmias
* Congestive heart failure (NYHA IV)
* Increased risk of bleeding
* Active internal bleeding or history of hemorrhagic diathesis
* History of TIA, ischemic or hemorrhagic stroke
* Intracranial neoplasm, aneurysm and arteriovenous malformation
* INR > 1.5 at screening
* Platelets < 100,000/ml
* Anemia (Hb < 10 g/dl) at screening
* One or more doses of a thienopyridine 5 d or less before PCI
* Oral anticoagulation which cannot be safely discontinued for the duration of the study
* One or more doses of a thienopyridine 5 d or less before PCI
* Treatment within the last 30 d with an investigational drug or are presently enrolled in another drug or device study
* Women who are known to be pregnant, have given birth within the past 90 d, or are breast-feeding
* Concomitant medical illness that in the opinion of the investigator is associated with reduced survival over the expected treatment period
* Known severe hepatic dysfunction
* Any condition associated with poor treatment compliance, including alcoholism, mental illness, or drug dependence
* Intolerance of or allergy to aspirin, ticlopidine, or clopidogrel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assessment of endothelial function (FMD) via high-resolution ultrasound (Sonoline G50, 12 MHz linear array transducer, Siemens, Germany) by experienced sonographer | baseline and after 3 months
  The primary endpoint is the change of endothelial function given in % from baseline to 3 months after therapy with prasugrel versus clopidogrel.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Rudolph, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- Cardiology, University Hospital of Cologne, Cologne, Germany